CLINICAL TRIAL: NCT00845143
Title: Vibration Response Imaging (VRI) in the Preoperative Management in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Ralf Eberhardt, MD, Thoraxklinik, University of Heidelberg
Other Study IDs: 003 HD
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Non-Small Cell Lung Cancer; Lung Function
Keywords: Non-small cell lung cancer; surgery; lung function
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the correlation of the predicted post-operative lung function with the observed post-operative lung function (FEV1 and DLCO) in patients who underwent surgical resection (FEV1 = Forced expiratory volume in 1-second. DLCO = Diffusion capacity for carbon monoxide. ppo = predicted postoperative.)and versus the gold standard QRRVP (Quantitative Radionuclide Study of Regional Lung Ventilation and Perfusion)

DETAILED DESCRIPTION:
The current standard lung function test uses radioisotopes (materials that produce radiation) injected in a vein and breathed into the lungs, which can show images of the function of the lungs.

The VRI system uses pressure sensors that act like electronic stethoscopes (tools used by doctors to listen to the heart and other sounds in the body). These sensors can record the energy (vibrations) created by the airflow in the lungs during the breathing process, which can then be visually imaged.

Before you can start this study, there will be a screening evaluation. The study doctor will review your medical record to find out if you are eligible to take part in this study. Information that will be viewed will include whether you have a skin lesion that might interfere with sensor placement, whether you have a cardiac pacemaker, and/or pregnancy test results. The study doctor will review with you the other types of information that will be viewed from your medical record to find out if you are eligible to take part in this study. For women who are able to have children, if you do not have a negative pregnancy test result in your medical record, you will not be able to take part in this study.

If you are found to be eligible and you agree to take part in this study, you will have a lung function test with the VRI system immediately before or after the standard lung function test. To perform the VRI test, you will be asked to remove your shirt and put on a garment to cover the front of your body. You will also be asked to remove your jewelry and other body accessories. You will then be asked to sit on a backless chair, and you will be instructed how to sit with the proper posture and breathe correctly for this test.

Before recording starts, the sensors will be cleaned and then placed on your back. You will be instructed to breathe deeply for up to 12 seconds (about 2-3 times), and the vibration responses will be recorded. You will have a total of 3 recording sessions, one after the other. Once all the recording is done, the sensors will be removed. The VRI image of the vibrations will then be examined by the operator in order to check the quality of the image.

The signals recorded from the sensors will be transferred to a computer so that researchers can study the images. The results of the recordings will be compared with the standard lung function test results. This will help researchers learn the level of accuracy of the VRI system in predicting how the lungs will function after surgery.

You will not be told of the results from the VRI testing because the results will not be used to diagnose your medical condition, nor will any medical decisions be made based on the VRI results. The VRI system is only used for investigational purposes in this study and will not replace the current diagnostic methods.

If you undergo surgery, as part of your standard care, you will also return to the clinic for standard tests to check your lung function 4-12 weeks and 4-12 months after your surgery. Researchers will compare your pre-surgery test results (both the standard test results and the VRI results) with the results of the tests after surgery (standard tests) to learn the level of accuracy of the VRI system in predicting how the lungs will function after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to read, understand, and provide written Informed Consent, and
2. Male or Female in the age range 18-90 years, and
3. Referred to perform QRRVP test for pre lung surgery evaluation due to lung cancer or other intrathoracic malignancy, and
4. BMI (body mass index) equal to or greater than 19

Exclusion Criteria:

1. Chest wall deformation, or
2. Spine deformation (including severe scoliosis), or
3. Hirsutism on back, or
4. Potentially contagious skin lesion on the back, or
5. Skin lesion that would interfere with sensor placement, or
6. Cardiac pacemaker or implantable defibrillator
7. Pregnancy (all women of childbearing age must have a negative pregnancy test before beginning the study) or breast feeding

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
lung function testing diffusion capacity VRI | pre- 6 weeks post and 3 month postoperative

REFERENCES:
- [Background] Yigla M, Gat M, Meyer JJ, Friedman PJ, Maher TM, Madison JM. Vibration response imaging technology in healthy subjects. AJR Am J Roentgenol. 2008 Sep;191(3):845-52. doi: 10.2214/AJR.07.3151. PMID 18716118
- [Background] Benditt JO. Surgical therapies for chronic obstructive pulmonary disease. Respir Care. 2004 Jan;49(1):53-61; discussion 61-3. PMID 14733622
- [Background] Kristersson S, Lindell SE, Svanberg L. Prediction of pulmonary function loss due to pneumonectomy using 133 Xe-radiospirometry. Chest. 1972 Dec;62(6):694-8. doi: 10.1378/chest.62.6.694. No abstract available. PMID 4635418
- [Result] Guntupalli KK, Reddy RM, Loutfi RH, Alapat PM, Bandi VD, Hanania NA. Evaluation of obstructive lung disease with vibration response imaging. J Asthma. 2008 Dec;45(10):923-30. doi: 10.1080/02770900802395496. PMID 19085584